CLINICAL TRIAL: NCT03529721
Title: Effect of Zumba Dance on Premenstrual Tension:8 Weeks Randomized Controlled Trial
Brief Title: Effect of Zumba Dance on Premenstrual Tension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zumba dance
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Premenstrual Tension
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zumba dance group (Experimental): females in this group will be instructed to engage into12 classes of 60-minute Zumba® fitness over an 8-week period of continuous dance movements to Latin music with varying intensity level throughout the sessions. Each session will be initiated with low-intensity movements for the ﬁrst 5 min, followed by an increasing intensity throughout the workout. At the end of the training session, the intensity will be gradually reduced.
  Interventions: Other: zumba dance fitness
- non zumba dance group (Placebo Comparator): the control group will be required to carry on doing their normal daily activities throughout the 8-week period.
  Interventions: Other: non zumba dance

INTERVENTIONS:
Other: zumba dance fitness — females in this group will be instructed to engage into12 classes of 60-minute Zumba® fitness over an 8-week period of continuous dance movements to Latin music with varying intensity level throughout the sessions. Each session will be initiated with low-intensity movements for the ﬁrst 5 min, followed by an increasing intensity throughout the workout. At the end of the training session, the intensity will be gradually reduced.
  Arms: zumba dance group
Other: non zumba dance — participants in this group will be doing their normal daily activities throughout the 8-week period.
  Other Names: control group
  Arms: non zumba dance group

SUMMARY:
Each female sets her experience of 47 manifestations on a 6 point scale separately for the premenstrual, menstrual and intermenstrual phases of her latest and worst menstrual cycle. Daily Symptoms Report will be filled at the start and at end of the study (before and after performing swimming exercise) Females in group I will be instructed to engage into 12 classes of 60-minute Zumba® fitness over an 8-week period.

DETAILED DESCRIPTION:
Each female sets her experience of 47 manifestations on a 6 point scale separately for the premenstrual, menstrual and intermenstrual phases of her latest and worst menstrual cycle. Daily Symptoms Report will be filled at the start and at end of the study (before and after performing swimming exercise) Females in group I will be instructed to engage into 12 classes of 60-minute Zumba® fitness over an 8-week period Each class was one hour in length and a recovery period of at least 48 hours will be taken between classes. The Zumba® fitness scheduling of sessions will be self-selected by the participants. The Zumba sessions will be conducted at a ﬁtness center (SAMIA ALLOUBA gym and fitness center) and will consist of continuous dance movements to Latin music with varying intensity level throughout the sessions. Each session will be initiated with low-intensity movements for the ﬁrst 5 min, followed by an increasing intensity throughout the workout. At the end of the training session, the intensity will be gradually reduced. The Zumba sessions will be supervised by three certiﬁed Zumba instructors, each responsible for regular sessions per week.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-25 years.
2. BMI :18-25 kg/m2.
3. A regular menstrual cycle of 23-35 days duration.
4. No previous practice of Zumba.
5. Free from musculoskeletal injury.
6. All women did not use oral contraceptive pills or any psychotropic agents.

Exclusion Criteria:

1. Pregnancy.
2. Metabolic/cardiorespiratory contraindications to physical exercise.
3. Cigarette smokers.
4. Recovering from a major injury or illness; or using anti-inflammatory, hyperlipidemia or hypertension medication.
5. any abnormality in ovulation or those with pelvic inflammatory diseases (PID) or a history of endometriosis.
6. Women with endocrine abnormality as diabetes mellitus, thyroid, pituitary, or ovarian disorders.
7. Women who are taking any hormonal drugs or drugs that affect hormones as antidepressant drugs during the preceding three months before the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Premenstrual distress questionnaire | 3 months after start of zumba dance fitness.
  47 manifestations on a 6 point scale separately for the premenstrual, menstrual and intermenstrual phases of her latest and worst menstrual cycle. Daily Symptoms Report will be filled at the start and at end of the study (before and after performing zumba dance fitness)

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Bahgat Gym and Spa, Cairo, Egypt